CLINICAL TRIAL: NCT03097926
Title: Prospective Randomized Trial of Duodenal Switch With a Standard Versus Long Alimentary Limb.
Brief Title: Duodenal Switch With a Standard Versus Long Alimentary Limb
Acronym: Long_limb_DS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Laurent Biertho, Clinical Professor, Laval University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DS long Limb
Record Dates: First submitted 2017-01-02; First posted 2017-03-31 (Actual); Last update posted 2018-03-27 (Actual); Status verified 2018-03

CONDITIONS: Obesity, Morbid; Bariatric Surgery Candidate; Metabolism Disorder
MeSH Terms: conditions — Obesity, Morbid; Metabolic Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard BPD-DS (Active Comparator): Standard BPD-DS with a 250-cm alimentary limb and 100-cm common channel
  Interventions: Procedure: Long alimentary limb BPD-DS
- Long alimentary limb BPD-DS (Experimental): BPD-DS with a 100-cm common channel, a 100-cm biliary limb, the remaining bowel as the strict alimentary channel
  Interventions: Procedure: Long alimentary limb BPD-DS

INTERVENTIONS:
Procedure: Long alimentary limb BPD-DS — BPD-DS with a long strict alimentary limb and a 100-cm common channel.

SUMMARY:
The aim of this study was to determine if Biliopancreatic Diversion with Duodenal Switch (BPD-DS) with a longer strict alimentary limb at the expense of a shorter biliopancreatic limb will offer significant weight lost, but with lesser gastrointestinal complaints, protein deficiency, vitamin and trace element deficit compared to standard BPD-DS.

DETAILED DESCRIPTION:
This two-group, randomized, single-blind pilot study is conducted in a university-affiliated tertiary care center. The study protocol was approved by our ethic committee. Enrollment and randomization of the patients occurred between May 20163 and June 2015. Patients are undergoing follow-up evaluation. Patients were initially referred to our center for a bariatric surgery evaluation. Eligible patients were 18 years of age or older and met the criteria for a laparoscopic biliopancreatic diversion. Patients were excluded if they had a BMI ≥ 50 mg/m², a pacemaker, cirrhosis or if they were planing pregnancy in the next 2 years. Each patient was required to provide written informed consent. Patients were randomly assigned in a 1:1 ratio to undergo a standard biliopancreatic diversion (control group) or a modified biliopancreatic diversion with a longer strict alimentary limb (study group). A sealed envelope with the assignation was given to the surgeon in the operation room just before the procedure. Patients are followed every 6 months after surgery, up to 24-months for clinical evaluation, resolution of comorbidities, evaluation of side-effects, quality of life, bioimpedance testing and bloodwork.

ELIGIBILITY:
Inclusion Criteria:

* Candidates for a biliopancreatic diversion, BMI above 35 with comorbidities or above 40 without comorbidities

Exclusion Criteria:

* BMI ≥ 50 mg/m², pacemaker, cirrhosis or planning pregnancy in the next 2 years, hypoalbuminemia, irritable bowel syndrome.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2013-05; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Total weight change | 6, 12, 18, 24 months
  Changes in total body weight, in kg, from baseline

SECONDARY OUTCOMES:
Changes in Gastro-intestinal side-effects scores | 6,12,18,24 months
  Gastro-intestinal symptoms assessed by measuring changes in GI Score
Changes in Quality of life | 6, 12, 18, 24 months
  Measure of Quality of life using Short-Form 36

OTHER OUTCOMES:
Resolution of Type 2 Diabetes | 6,12,18,24 months
  Resolution rate of T2DM (based on normalized HbA1c without medication)
Resolution of Hypertension | 6,12,18,24 months
  Resolution rate of hypertension, base on normalized blood pressure without medication
Resolution of dyslipidemia | 6,12,18,24 months
  Percentage of patients with normalized cholesterol without medication
Resolution of sleep apnea | 6,12,18,24 months
  Percentage of patients with normalized sleep apnea testing without airway support

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Biertho, MD, Principal Investigator — Quebec Heart and Lung Institute

IPD SHARING:
Plan to Share IPD: Undecided
Publication in peer-reviewed journal

REFERENCES:
- [Derived] Malo FC, Marion A, Rioux A, Lebel S, Hould F, Julien F, Marceau S, Lescelleur O, Lafortune A, Bouvet-Bouchard L, Biertho L. Long Alimentary Limb Duodenal Switch (LADS): an Exploratory Randomized Trial, Results at 2 Years. Obes Surg. 2020 Dec;30(12):5047-5058. doi: 10.1007/s11695-020-04968-5. Epub 2020 Sep 17. PMID 32940866